CLINICAL TRIAL: NCT05839509
Title: A Phase 2 Clinical Trial of GH001 in Patients with Bipolar II Disorder and a Current Major Depressive Episode
Brief Title: Phase 2 Clinical Trial of GH001 in Bipolar II Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment of this patient population was more challenging than anticipated. The sponsor concluded that a sufficient amount of patients have completed the trial to demonstrate proof of concept in this patient population.
Sponsor: GH Research Ireland Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GH001-BD-202
Record Dates: First submitted 2023-04-20; First posted 2023-05-03 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Bipolar II Disorder
Keywords: Depression; Bipolar Disorder; 5-Methoxy-N,N-Dimethyltryptamine; 5-MeO-DMT; Mebufotenin
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Methoxydimethyltryptamines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GH001 Individualized Dosing Regimen (Experimental): GH001 (Mebufotenin, 5-Methoxy-N,N-Dimethyltryptamine) is administered via inhalation, as an IDR consisting of up to 3 increasing doses of GH001 (6 mg, 12 mg, and 18 mg), on a single day. The second and third doses are only administered if the patient did not achieve intense psychoactive effects (a peak experience [PE]) at the previously administered dose.
  Interventions: Drug: GH001

INTERVENTIONS:
Drug: GH001 — GH001 administered via inhalation
  Other Names: 5-Methoxy-N,N-Dimethyltryptamine; 5-MeO-DMT; Mebufotenin

SUMMARY:
This study is a multicenter, open-label, single-arm Phase 2 clinical trial. Approximately 15 participants with clinically diagnosed bipolar disorder (BD) type II and experiencing a current episode of depression will be included in this study. The participants will receive an individualized dosing regimen (IDR) with at least one and up to three doses of GH001 administered within a single day.

ELIGIBILITY:
Inclusion Criteria:

* Is male or female and in the age range between 18 and 64 years (inclusive) at screening
* Has a body mass index (BMI) in the range of 18.5 and 35 kg/m2 (inclusive) at screening
* Meets the trial criteria for bipolar II disorder and is experiencing a major depressive episode, as assessed by a trial psychiatrist or registered clinical psychologist

Exclusion Criteria:

* Has bipolar II disorder with rapid cycling (four or more episodes of hypomania or depressive episodes in previous 12-month period)
* Has, based on history, psychiatric assessment, and evaluation of the MINI, a current or prior diagnosis of bipolar I disorder, a manic episode, a psychotic disorder, MDD or other mood disorder with psychotic features, obsessive compulsive disorder, PTSD, autism spectrum disorder, borderline personality disorder, schizophrenia, delusional disorder, paranoid personality disorder, schizoaffective disorder, clinically significant intellectual disability, or any other psychiatric comorbidity that renders the patient unsuitable for the trial according to the investigator's judgment
* Has one or more first degree relatives with a current or previously diagnosed psychotic disorder, bipolar I disorder or MDD with psychotic features
* Has taken prohibited medication or prohibited dietary supplements within the specified timeframe prior to dosing
* Has previously experienced a significant adverse reaction to a hallucinogenic or psychedelic drug according to the investigator's judgment
* Has a clinically significant abnormality in physical examination, vital signs, ECG, or clinical laboratory parameters which renders the patient unsuitable for the trial according to the investigator's judgment

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
The anti-depressive effects of GH001 evaluated by the change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) assessed at Day 7 | From Baseline to Day 7
  The MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. A higher MADRS score indicates more severe depression, and each item is scored from 0 to 6. The overall score ranges from 0 to 60.

CONTACTS AND LOCATIONS:
Locations (7):
- Germany (3):
  - Investigational Site, Dresden
  - Investigational Site, Frankfurt
  - Investigational Site, Münster
- Netherlands (2):
  - Investigational Site, Leiden
  - Investigational Site, Maastricht
- United Kingdom (2):
  - Investigational Site, London
  - Investigation Site, Oxford

IPD SHARING:
Plan to Share IPD: No